CLINICAL TRIAL: NCT01892527
Title: A Single-Arm Phase II Study of Tivantinib (ARQ 197) Plus Cetuximab in EGFR Inhibitor-Resistant MET High Subjects With Locally Advanced or Metastatic Colorectal Cancer With Wild-Type KRAS
Brief Title: Study of Tivantinib (ARQ 197) Plus Cetuximab in EGFR Inhibitor-Resistant MET High Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, Medical Doctor - Oncologist, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2012-001
Record Dates: First submitted 2013-05-06; First posted 2013-07-04 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer Metastatic; C-met Overexpression
Keywords: Colorectal Cancer Metastatic; wild type KRAS; C-met overexpression; Tivantinib; Cetuximab
MeSH Terms: interventions — ARQ 197; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tivantinib plus Cetuximab (Experimental): Single arm
  Interventions: Drug: Tivantinib (ARQ197)

INTERVENTIONS:
Drug: Tivantinib (ARQ197) — Eligible subjects will be treated with tivantinib (ARQ 197) at a dose of 360 mg twice daily (a total daily dose of 720 mg) orally in a continuous manner and cetuximab (Erbitux) at a dose of 500 mg/mq i.v. every 2 weeks.
  Other Names: Cetuximab

SUMMARY:
This is a single-arm, Simon 2-stage, phase 2 clinical study conducted in subjects with advanced or metastatic colorectal cancer who have previously received ≥ 1 prior line of systemic therapies and are resistant to EGFR inhibitor (cetuximab or panitumumab).

This trial will be conducted to determine objective response rate (ORR), progression-free survival (PFS) and overall-survival (OS) of cetuximab plus tivantinib in patients with wild-type KRAS CRC that is resistant to anti-EGFR antibody treatment (cetuximab or panitumumab) and shows overexpression of cMET.

DETAILED DESCRIPTION:
This is a single-arm, Simon 2-stage, phase 2 clinical study conducted in subjects with advanced or metastatic colorectal cancer who have received ≥1 prior line of systemic therapies and are resistant to EGFR inhibitor (cetuximab or panitumumab). Fresh tumor tissue is needed for the MET testing, thus a biopsy will be required to participate in this trial. In a minor percentage of subjects archival tumor tissue could be acceptable for this analysis.Eligible subjects will be treated with tivantinib (ARQ 197) at a dose of 360 mg twice daily (a total daily dose of 720 mg) orally in a continuous manner and cetuximab (Erbitux) at a dose of 500 mg/mq i.v. every 2 weeks. The overall treatment period will be divided into continuous 28 days cycles without treatment interruption. Disease status and tumor response will be assessed per modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 at screening (within 4 weeks before the first scheduled dose of study drug), in 8 weeks intervals while the subjects are on treatment or as clinically indicated until progression of disease, withdrawal of consent, death, or lost to follow-up. Tumor measurement will also be performed during the end of treatment visit if not done within the previous 8 weeks. Subjects with progressive disease at any time during the treatment period will discontinue study treatment. Subjects with stable disease (SD), complete response (CR) and partial response (PR) will stay on treatment until disease progression and/or unacceptable toxicity and/or withdrawal of consent is documented. CR and PR must be confirmed no sooner than 4 weeks after the initial observation. After discontinuation from study treatment during the follow-up period, survival status will be obtained by phone every 3 months until the subject dies, withdraws consent from study, or is lost to follow-up, for a maximum of 12 months.

ELIGIBILITY:
Inclusion Criteria:Subjects must satisfy all of the following criteria to be included in the study:

1. Subjects with surgically unresectable locally advanced or metastatic disease who have received ≥ 1 prior line of systemic therapies for advanced or metastatic disease. The last treatment regimen must include EGFR inhibitor (cetuximab or panitumumab) on which the patient had a best response as CR or PR or SD, and must have either progressed on or after EGFR inhibitor based therapy within 3 months before enrollment. Subjects must have radiologically documented disease progression prior to enrollment.
2. All subjects must express the wild-type form of the gene KRAS. Previously existing KRAS mutation status from an accredited local laboratory will be accepted.
3. Fresh tumor biopsy tissue must be available for molecular sequencing and biomarker expression in >70% of patients. If prior radiotherapy, tissue biopsy must be outside radiotherapy field. In a minor percentage of patients (<30%) archival tumor tissue could be considered acceptable for molecular sequencing and biomarker expression.
4. Patients must be MET High testing by IHC (IHC 2+ or 3+ in ≥50% of tumor cells) analyzed by Ventana Test Kit.
5. Measurable disease according to RECIST criteria, Version 1.1.
6. Male or female ≥ 18 years of age.
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
8. Resolution of any toxic effects of prior therapy to NCI CTCAE, Version 4.0, grade ≤ 1 (with the exception of alopecia and grade ≤ 2 neuropathy).
9. Adequate bone marrow, liver, and renal functions, defined as: Hemoglobin ≥ 9.0 g/dL (transfusion and/or growth factor support allowed).

   Absolute neutrophil count (ANC) ≥ 1.5 × 109/L. Platelet count ≥ 75 × 109/L. Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min. Alanine transaminase (ALT), and aspartate transaminase (AST) ≤ 2.5 x ULN in subjects with no liver metastasis and ≤ 5.0 x ULN in subjects with liver metastasis. Total bilirubin ≤ 1.5 x ULN (≤ 4 x ULN and direct bilirubin ≤ 1.5 x ULN is acceptable for subjects with Gilbert's syndrome).
10. Male and female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received. 11. All female subjects of childbearing potential must each have a negative pregnancy test (serum or urine) result before initiating study treatment.

12. Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an IEC- or IRB-approved ICF (including HIPAA authorization, if applicable) before performance of any study-specific procedures or tests.

Exclusion Criteria:

Subjects who meet any of the following criteria will be disqualified from entering the study:

1. History of malignancy other than CRC, unless there is an exception that the malignancy has been cured and no tumor- specific treatment for the malignancy has been administered within the 3 years prior to initiation of study treatment (subjects with a history of basal cell carcinoma or benign tumor of cervix can be enrolled if diagnosis and treatment occurred < 3 years prior to enrollment).
2. Anticipation of need for a major surgical procedure or radiation therapy (RT) during the study.
3. Treatment with chemotherapy, radiotherapy, surgery, immunotherapy, biological therapy, or any other investigational anticancer agent within 3 weeks prior to start of study treatment.
4. History of cardiac disease: Congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD); Previously diagnosed bradycardia (subjects with asymptomatic bradycardia and hear rate above 50 bpm are allowed) or other cardiac arrhythmia defined as ≥Grade 2 or higher according to NCI CTCAE, version 4.0, or uncontrolled hypertension; myocardial infarction that occurred within 6 months prior to start of study treatment (myocardial infarction that occurred > 6 months prior the start of study treatment is permitted).
5. Malabsorption syndrome, chronic diarrhea (lasting > 4 weeks), inflammatory bowel disease, or partial bowel obstruction.
6. Known metastatic brain or meningeal tumors, unless the subject is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of first dose of study treatment, and is clinically stable (no concomitant therapy, including supportive therapy with steroids or anticonvulsant medications) with respect to the tumor at the time of first dose of study treatment.
7. Uncontrolled seizure disorder, spinal cord compression, or carcinomatous meningitis.
8. Pericardial or pleural effusion (requiring drainage) or pericardial involvement with the tumor. Subjects with minimal pleural effusion may be eligible upon request by Investigator and approval by Sponsor.
9. Clinically significant active infection that requires antibiotic therapy.
10. Previous administration of any MET inhibitor (including tivantinib) or EGFR inhibitor (except cetuximab or panitumumab).
11. Substance abuse or medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the subject's participation in the clinical trial or evaluation of the clinical trial results.
12. Any condition that is unstable or that could jeopardize the safety of the subject and the subject's protocol compliance.
13. Inability to swallow oral medications.
14. Pregnant or nursing females.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Study of Tivantinib (ARQ 197) plus Cetuximab in EGFR inhibitor-Resistant MET High Subjects with Locally Advanced or Metastatic Colorectal Cancer with Wild-Type KRAS | 36 months
  To determine objective response rate (ORR).

SECONDARY OUTCOMES:
Tivantinib (ARQ 197) plus Cetuximab in EGFR inhibitor-Resistant MET High Subjects | 36months
  To estimate progression-free survival (PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenza Rimassa, MD, Study Chair — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy